CLINICAL TRIAL: NCT03177746
Title: The Safety of Dapoxetine/Tadalafil Combination Therapy in Treatment of Men With Premature Ejaculation and Erectile Dysfunction
Brief Title: The Safety of Dapoxetine/Tadalafil Combination Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-10.16
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Premature Ejaculation; Erectile Dysfunction; Safety Issues
MeSH Terms: conditions — Premature Ejaculation; Erectile Dysfunction | interventions — dapoxetine; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapoxetine/Tadalafil 30/20 mg film coated tablet (Experimental)
  Interventions: Drug: Dapoxetine/Tadalafil 30/20 mg film coated tablet

INTERVENTIONS:
Drug: Dapoxetine/Tadalafil 30/20 mg film coated tablet — During 4-weeks treatment period, patients will take one Dapoxetine/Tadalafil 30/20 mg film coated tablet 1-3 hours before sexual intercourse.
  Study drug should not be used more than 1 tablet every 24 hours during the treatment.
  Other Names: Tada Plus

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Dapoxetine/Tadalafil 30/20 mg film-coated tablet in the treatment of men with premature ejaculation and erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old men,
* Participants must be heterosexual males and in a stable monogamous sexual relationship with a female partner for at least 6 months and will continue throughout the study,
* Clinical diagnosis of erectile dysfunction, IIEF score ≤21,
* Premature Ejaculation Diagnostic Tool (PEDT) score must be ≥11
* Patients with life-long PE and acquired PE according to the description of International Society for Sexual Medicine (ISSM) ,
* The patient and his partner must have sexual intercourse twice a week for the duration of the study,
* Commitment to comply with the study protocol,
* Patients who sign informed consent form (ICF).

Exclusion Criteria:

* History of medical events such as surgical interventions or neurologic conditions (e.g., multiple sclerosis), trauma, or infections that are associated with the development of symptoms of premature ejaculation (PE) and considered a potential cause of PE,
* Having genital abnormalities, except penile curvature unless not prevent sexual intercourse,
* Developed erectile dysfunction or premature ejaculation due to drug use or quit taking drugs,
* Any conditions that prevent sexual intercourse with partners
* History of epilepsy,
* Severe renal insufficiency,
* Liver disease,
* History of in last 6 months stroke, myocard infarction, cardiac insufficiency (New York Cardiovascular Associates (NYCA) phase II-IV), atrioventricular block or message disorder such as sick sinus syndrome, severe ischemic cardiac disease, syncope, unstable angina, life-threatening arrhythmia or hypotension,
* Non-Arteritic Anterior ischemic optic neuropathy,
* Patients who are not eligible to have sexual intercourse due to existing health problems,
* Autonomic neuropathy, retinitis pigmentosa, blood diseases, active peptic ulcer, abnormalities in ECG, severe systemic disease that cannot be controlled,
* Systolic/Diastolic blood pressure at rest <90/50 mmHg and 170/100 mmHg<
* History of allergy to Selective Serotonin Reuptake Inhibitor (SSRI) and phosphodiesterase inhibitor drugs,
* Continuing to use or quitted in last 3 months of Monoamine oxidase inhibitor (MAOI), Thioridazine, Serotonin Reuptake Inhibitor (SSRI), Selective-norepinephrine Reuptake Inhibitor (SNRI), Serotonergic drug/herbal product, tricyclic antidepressant and atypical antipsychotic drugs,
* Use of nitrates, alfa blockers, vasodilators, ketoconazole, itraconazole, ritonavir, saquinavir, telithromycin, nefazodone, nelfinavir, atazanavir, cimetidine, erythromycin, clarithromycin, fluconazole, amprenavir, fosamprenavir, aprepitant, verapamil, diltiazem, any kind of vasodilator, antiplatelet, anticoagulant, dapoxetine, phosphodiesterase 5 inhibitor, alcohol and stimulant drug,
* Patients on a different therapy (behavioral therapy or other drugs that are applied locally) for PE treatment
* During the study, the possibility of taking medication which may affect the study drug's pharmacokinetic/pharmacodynamic properties
* Patients who are defining symptoms of prostatitis clinically
* Thyroid hormone disorders

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since drug is indicated in men, study population will consist of men.
Enrollment: 40 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2023-01-14 (Estimated); Study Completion 2023-10-14 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety of study drug | 4 weeks
  Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Evaluation of change in Intra-vaginal Ejaculation Latency Time (IELT) compared to baseline | 4 weeks
  Intra-vaginal ejaculation latency time difference of one minute or more will be considered as efficient.
Evaluation of IIEF-15 (International Index of Erectile Function) score compared to baseline | 4 weeks
  Increase in IIEF score will be considered as efficacy.
Evaluation of premature ejaculation symptom scores compared to baseline | 4 weeks
  Increase in IIEF scores will be considered as efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Okmeydanı Training and Research Hospital Urology Dep., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided